CLINICAL TRIAL: NCT06612775
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety, Tolerability, and Efficacy of CB03-154 as Adjunctive Therapy in Focal Epilepsy
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of CB03-154 in Adult Patients With Focal Epilepsy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB03-154-EP201
Record Dates: First submitted 2024-09-19; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CB03-154 5mg and Placebo 15mg (Experimental): Participants will receive CB03-154 5mg and Placebo 15mg orally once daily for 12 weeks.
  Interventions: Drug: Test drug CB03-154 5mg group
- CB03-154 10mg and Placebo 10mg (Experimental): Participants will receive CB03-154 10mg and Placebo 10mg orally once daily for 12 weeks.
  Interventions: Drug: Test drug CB03-154 10mg group
- CB03-154 20mg (Experimental): Participants will receive CB03-154 20mg orally once daily for 12 weeks.
  Interventions: Drug: Test drug CB03-154 20mg group
- Placebo 20mg (Placebo Comparator): Participants will receive Placebo 20mg orally once daily for 12 weeks.
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Test drug CB03-154 5mg group — CB03-154 tablet (5mg/tablet) once daily.
  Arms: CB03-154 5mg and Placebo 15mg
Drug: Test drug CB03-154 10mg group — Two CB03-154 tablets (5mg/tablet) once daily.
  Arms: CB03-154 10mg and Placebo 10mg
Drug: Test drug CB03-154 20mg group — Four CB03-154 tablets (5mg/tablet) once daily.
  Arms: CB03-154 20mg
Drug: Placebo group — Four Placebo tablets once daily.
  Arms: Placebo 20mg

SUMMARY:
CB03-154 is an investigational drug developed by Shanghai Zhimeng Biopharma Inc. for the treatment of Focal Epilepsy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of CB03-154 on focal seizure frequency by comparing with placebo, see how safe the study drug is and assess how well it is tolerated after dosing in adults with focal epilepsy taking 1 to 3 AEDs in the double-blind trial. The study will also test the 50% response rates of the study drug and see how it is taken up and eliminated by the body. An additional part of the study is to look how will the study drug influence the trends of frequency and seizure severity in the double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of the subjects or his/her authorized representative be fully informed of the nature and risks of the study and give informed consent in writing prior to entering the study.
2. Male and female aged 18 to 70 years, inclusive.
3. 18.0 kg/m2 ≤BMI ≤ 34.0 kg/m2.
4. Diagnosis (≥2 years) of focal epilepsy according to the International League Against Epilepsy [ILAE] Classification of Epilepsy (2017).
5. Prior neuroimaging within the last 5 years and documentation are available to rule out progressive structural central nervous system abnormalities at the time of the diagnosis of epilepsy.
6. Treatment with a stable dose of 1 to 3 allowable current AEDs for at least one month prior to screening, during baseline, and throughout the duration of the DBP.
7. Prior to screening and during baseline period, subjects must have at least 6 focal seizures without status epilepticus, with or without focal to bilateral tonic-clonic.
8. If a female, must be:

   * Postmenopausal, defined as amenorrhea for at least 12 months, and confirmed by blood follicle stimulating hormone (FSH) at Screening, OR
   * Surgically sterile with a documented hysterectomy, partial hysterectomy, bilateral oophorectomy, or bilateral tubal ligation at least 6 months prior to Screening, OR
   * If of child-bearing potential, heterosexually active females with male partners must be using an acceptable and highly effective method of contraception at least one menstrual cycle before first study drug administration and continuing until at least 3 months after the last dose of the study drug. If a female subject is abstinent, she must agree to use an acceptable and highly effective form of birth control as above once she becomes heterosexually active during the study.
9. If a female of child-bearing potential, must have a negative pregnancy test result at Screening and Check-in.
10. If a male, if heterosexually sexually active with a female partner of child-bearing potential and has not had a vasectomy, must agree to use a highly effective method of contraception and deemed appropriate by the Investigator and must not donate sperm during the study and for 3 months after the last dose of study drug.
11. Able to keep accurate seizure diaries.

Exclusion Criteria:

1. Subject has had documented previous EEGs indicating other patterns of epilepsy besides the focal epilepsy prior to dosing the study drug.
2. Subject has seizures secondary to drugs or alcohol use, ongoing infection, metabolic diseases or progressive central nervous system diseases or lesions at the investigator's assessments.
3. Subject has the history of pseudo seizures, conversion disorders, or other non-epileptic seizure conditions, or other non-epileptic ictal events that could be confused with seizures at the investigator's discretion and/or EEG evidence.
4. Subject has the presence or previous history of Lennox-Gastaut syndrome, some other related syndrome or evidence of both focal and generalized epilepsy at investigator's decisions.
5. Subject has the history of status epilepticus within 6 months prior to screening.
6. Subject has only uncountably repetitive seizures occurring within 6 months prior to screening.
7. Subject has the history of neurosurgery for seizures <1 year prior to enrolment, or radiosurgery <2 years prior to enrolment. Subjects has the implantment and activation of vagus nerve stimulation (VNS), deep brain stimulation (DBS), or other neurostimulation for epilepsy treatment <1 year prior to enrolment, or with stimulation parameters that have been stable for <3 months prior to enrolment, or with anticipated left battery lifetime shorter than trial duration.
8. Subject has any of the following findings will be excluded:

   * A history or family history of unexplained syncope;
   * A history of presence of long QT syndrome; QTcF > 450 msec prior to first dose of the study drug; a family history of long QT syndromes or sudden death of unknown cause;
   * Bundle branch blocks or atrioventricular or other conduction abnormalities that are clinically significant according to the Investigator and/or with a PR interval ≥220ms, or HR<50bpm at rest in ECGs or vital signs, prior to first dose of the study drug;
   * A history of venous thrombosis, or a history or presence of medical conditions indicating unresolved high risks of thrombophilia or hypercoagulability including but not limited to protein C deficiency, protein S deficiency, antithrombin deficiency, antiphospholipid syndrome, Budd-Chiari syndrome, myeloproliferative neoplasm including Chronic myeloid leukemia (CML), polycythemia vera (PV), essential thrombocythemia (ET) and primary myelofibrosis (PMF), autoimmune diseases (especially systemic lupus erythematosus (SLE) or antiphospholipid syndrome or vasculitis), nephrotic syndrome, paroxysmal nocturnal hemoglobinuria, uncured malignancy, unstoppable estrogen containing oral or injection contraception or hormone replacement therapy, postpartum period within 2 months, or other medical conditions at the investigator and the medical monitor's judgements;
   * Venous ultrasound examinations on bilateral lower extremes indicating DVT;
   * > 2.0 Upper limit of normal (ULN) of blood D-Dimer, or >1.5 Upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma-glutamyl transpeptidase (GGT), amylase (AMY) prior to first dose of the study drug. If subject has >ULN of above laboratory tests that does not meet the exclusion limit at screening, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase at the investigator's and/or the medical monitor's judgments;
   * The estimated glomerular filtration rate (eGFR) at screening is <60mL/min and the calculated result of female is ×0.85.
9. Subject has any clinically significant abnormalities on physical examination, vital signs, laboratory tests or ECG prior to first dose of the study drug which could jeopardize or would compromise the subject's safety or ability to participate in this study as deemed by the Investigator and the Medical monitor.
10. Subject has the history or presence of significant medical or surgical condition including but not limited to cardiac, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, psychiatric disease, or history of cancer within the past 2 years, with the exception of appropriately treated basal cell or squamous cell carcinoma, or any condition which could jeopardize or would compromise the subject's safety or ability to participate in this study in the opinion of the investigator and/or the medical monitor at enrolment.
11. Subject with active pathogen infections or carrier including but not limited to testing positive at Screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody or syphilis.
12. Subject has schizophrenia and other psychotic disorders, or active suicidal plan/intent in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening, or a history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt) within 2 years prior to enrolment, or more than 1 lifetime suicide attempt.
13. Subject ever used vigabatrin without no vigabatrin-related visual field abnormalities confirmed by examination within the past 6 months at screening (concomitant use of vigabatrin is not allowed).
14. If felbamate will be a concomitant AED during study, the subject must be on felbamate for at least 2 years, and with a stable dose for at least 2 months prior to screening and without planned changes of the dose during the study. Subject must not have a history of white blood cell (WBC) count below 3000/μL (3.00 *109/L), platelets below 75,000/mm3 (75*109/L), liver function tests above 1.5 times the ULN, or other indication of hepatic or bone marrow dysfunction while receiving felbamate. If felbamate was ever used before, it must have been discontinued for at least 2 months prior to screening.
15. Subject has taken other (non-AED) prescription, nonprescription, dietary (e.g., grapefruit or passion fruit), or herbal products that are potent inducers or strong or moderately inhibitors of the CYP3A4 pathway for 2 weeks prior to the baseline.
16. Subject has received an investigational medicinal product within 3 months or within 10 half-lives of the drug (whichever is longer) or IMP of monoclonal antibodies, cytokines, growth factors, soluble receptors, other recombinant products, or fusion proteins within 6 months prior to the first dose of study drug.
17. Subject is known allergic or hypersensitive to any of excipients of CB03-154 tablet formulation.
18. Subject has had multiple drug allergies or a severe drug reaction to an AED(s), including dermatological, hematological, or organ toxicity reactions.
19. Subject has a history of indicated alcohol abuse or drug abuse at the investigator's decision during the 6 months prior to screening. Subject tested positive for substance abuse at screening or check-in.
20. Female subject who is pregnant or in the postpartum period within 2 months or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of CB03-154 compared to placebo on focal seizure frequency in adults with focal epilepsy taking 1 to 3 AEDs in the double-blind period (DBP). | From baseline to the entire period of double-blind period, assessed up to 20 weeks.
  Median percent change (MPC) in monthly (28 days) focal seizure frequency from baseline to the entire period of DBP for CB03-154 versus placebo.
To assess the safety and tolerability by evaluating the frequency and severity of adverse events (AEs) /serious adverse events (SAEs) of CB03-154 in adults with focal epilepsy taking 1 to 3 AEDs in the DBP. | From the entire period of double-blind period of 12 weeks to the post-treatment follow-up period of 2 weeks(+7 days), assessed up to 17 weeks.
  Severity and frequency/incidence of associated AEs/serious adverse events (SAEs).

SECONDARY OUTCOMES:
To evaluate the 50% CB03-154 response rates in comparison to placebo in the DBP. | From baseline to the entire period of double-blind period, assessed up to 20 weeks.
  Proportion of responders, defined as experiencing ≥50% reduction in monthly (28 days) focal seizure frequency at baseline compared to the entire period of DBP.
To evaluate trends in focal seizure frequency over time in the DBP. | From baseline to the entire period of double-blind period, assessed up to 20 weeks.
  Percent change from baseline in weekly focal seizure frequency for each week of the DBP.
Maximum Plasma Concentration (Cmax). | On Day 7, Day 15, Day 29, and Day 85 in the period of double-blind period.
  For all subjects, blood will be collected on Day 7, Day 15, Day 29, and Day 85 in the period of double-blind period for plasma concentration measurement.
Use the Hamilton Depression Rating Scale (HAMD-17) to assess the effect of CB03-154 vs placebo on seizure severity and impact in adults with focal epilepsy taking 1 to 3 AEDs in the DBP. | In the entire period of double-blind period, assessed up to 12 weeks.
  To assess the change from baseline to the end of DBP in the Hamilton Depression Rating Scale (HAMD-17) total score during the DBP. The total score can better reflect the severity of depression, the lighter the illness, the lower the total score. A score above 24 was severe depression, 17 to 24 was moderate depression, 7 to 17 was mild depression, and a score below 7 was no depressive symptoms.
Clinical Global Impression of Change (CGI-C) scores during the DBP. | In the entire period of double-blind period, assessed up to 12 weeks.
  The CGI-C scale (National Institute of Mental Health [NIMH]) will be administered by a trained physician at selected visits as specified in schedule of assessments.
Patient Global Impression of Change (PGI-C) scores during the DBP. | In the entire period of double-blind period, assessed up to 12 weeks.
  The PGI-C scale (National Institute of Mental Health [NIMH]) will be provided to the patient for completion at selected visits as specified in in schedule of assessments.

IPD SHARING:
Plan to Share IPD: No